CLINICAL TRIAL: NCT04621981
Title: Sodium Bicarbonate Ringer's Solution Versus Normal Saline for Early Fluid Resuscitation in Patients With Sepsis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RIN005-R
Record Dates: First submitted 2020-11-01; First posted 2020-11-09 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Sepsis, Septic Shock
Keywords: Fluid Resuscitation, Crystalloid Solution
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — bicarbonated Ringer's solution; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Bicarbonate Ringer's Solution (Experimental): Intravenous drip, 500~1000ml per time. Infusion speed: 15ml/kg/h or according to guidelines or department routine.
  Interventions: Drug: Sodium Bicarbonate Ringer's Solution
- Normal Saline (Active Comparator): Intravenous drip, 500~1000ml per time. Dosage depends on age、weight and symptoms.
  Infusion speed: According to the department process or clinician's decision.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Sodium Bicarbonate Ringer's Solution — This group was treated with Sodium Bicarbonate Ringer's Solution.
  Other Names: Bicarbonated Ringer's solution
  Arms: Sodium Bicarbonate Ringer's Solution
Drug: Normal Saline — This group was treated with normal saline.
  Other Names: physiological saline
  Arms: Normal Saline

SUMMARY:
At present, people still have different opinions on choosing which kind of crystalloid solution for patients with sepsis, and there is no unified standard yet. It is necessary to conduct systematic studies on comparison of different fluid resuscitation methods on the efficacy and safety of crystalloid solution for patients with sepsis. Therefore, this study focuses on the efficacy and safety of sodium bicarbonate Ringer's solution compared with normal saline.

DETAILED DESCRIPTION:
Sepsis and septic shock are clinical emergencies requiring immediate treatment and fluid resuscitation. Early effective fluid resuscitation can improve the prognosis of patients. So far, there is no perfect crystalloid solution. Normal saline is the most readily available and economical crystalline fluid for clinical resuscitation. It is isoosmotic and can meet the basic needs of patients in the early rehydration. But it lacks acid-base buffer system and potassium, calcium and magnesium ions, and the level of chloride ions is also significantly higher than that of plasma.

Sodium Bicarbonate Ringer's solution contains physiological levels of Na+(130mmol/L), K+(4mmol/L), Ca2+(1.5mmol/L), Mg2+(1mmol/L), HCO3-(28mmol/L) and Cl-(109mmol/L). It also has citric acid/ sodium citrate buffer system (Citrate3-1.3mmol/L), pH7.3, and osmotic pressure 276mOsm/L. It is the most similar solution to extracellular fluid.

Theoretically，Compared with normal saline, Sodium Bicarbonate Ringer's solution can maintain acid-base balance faster and better when restoring the microcirculation without affecting the level of chloride ion. Therefore we hypothesize that Sodium Bicarbonate Ringer's solution can promote the body to restore to acid-base balance more quickly, and improve organ function more significantly than normal saline.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as sepsis or septic shock according to the definition of Sepsis-3.0 with fluid resuscitation requirement;
* aged between 18 and 80, male or female;
* Signed informed Consent (with delay within 24 hours).

Exclusion Criteria:

* Patients with hypermagnesemia;
* Patients with hypothyroidism;
* Patients predicted to die or discharged within 24 hours after admission;
* Patients with previous history of mental illness, severe hepatic and renal insufficiency, severe cardiac disease, primary severe central nervous system lesions;
* Pregnant or breast-feeding women;
* Patients who have received cardiopulmonary resuscitation；
* Patients who participated in other clinical trials within 30 days;
* Patients have other conditions that are not appropriate for inclusion according to the researcher's judgment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2021-03-11 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Sequential Organ Failure Assessment(SOFA) value at 24h | 0 hours, 24 hours
  ΔSOFA=SOFA24h-SOFA0h

SECONDARY OUTCOMES:
Serum lactate clearance rate | 0 hours, 6 hours
  (Serum lactete0h-serum lactate6h)/serum lactate0h
The proportion of patients with serum lactate clearance rate>30% | 0 hours, 6 hours, 24 hours
  the proportion of patients whose serum lactate decrease by more than 30%
Changes in pH value over time, and the lowest pH value during hospitalization | 0 hours, 3 hours, 6 hours, 24 hours
  ΔpH=pH3h/6h/24h-pH0h, and the lowest pH value during hospitalization
Changes in base residue (BE value) over time | 0 hours, 3 hours, 6 hours, 24 hours
  ΔBE=BE3h/6h/24h-BE0h
Changes in serum bicarbonate(HCO3-) over time | 0 hours, 3 hours, 6 hours, 24 hours
  ΔHCO3-=HCO3-3h/6h/24h-HCO3-0h
The proportion of patients with hyperchloremia | 0 hours, 3 hours, 24 hours
  The proportion of patients with hyperchloremia at 3h and 24h.
Changes in SOFA score over time | 0 hours, 24 hours, 48 hours, 72 hours
  ΔSOFA=SOFA24h/48h/72h-SOFA0h
Changes in APACHEII score over time | 0 hours, 24 hours, 48 hours, 72 hours
  ΔAPACHEII=APACHEII24h/48h/72h-APACHEII0h
Mechanical ventilation time(h) | Within 7 days
  the length of mechanical ventilation time within 7 days
The proportion of patients receiving RRT | Within 7 days
  The proportion of patients receiving RRT within 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Lina Zhang, Principal Investigator — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China